CLINICAL TRIAL: NCT06023446
Title: Illuminating Glial Dysfunction in Alzheimer's Disease With Optical Coherence Tomography
Brief Title: Can (Optical Coherence Tomography) Pictures of the Retina Detect Alzheimer's Disease at Its Earliest Stages?
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1647468; K08AG080178 (NIH)
Record Dates: First submitted 2023-07-21; First posted 2023-09-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Amyloid; Retinal Muller Glial Cells; Optical Coherence Tomography; Glia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Dementia Alzheimer's: By clinical assessment, these participants will either be cognitively normal, or have mild cognitive impairment. They will enter the study having already completed some biomarker testing for Alzheimer's disease (e.g., amyloid PET, cerebrospinal fluid measurement amyloid and tau). In this group, the biomarker testing is positive/abnormal, indicating a pre-dementia stage of Alzheimer's disease. In the language of the 2018 NIA-AA Research Framework, these participants have A+ in their AT(N) biomarker profile, and are at clinical stage 1-3.
  Interventions: Diagnostic Test: Optical Coherence Tomography
- No Evidence of Alzheimer's: By clinical assessment, these participants will either be cognitively normal, or have mild cognitive impairment. They will enter the study having already completed some biomarker testing for Alzheimer's disease (e.g., amyloid PET, cerebrospinal fluid measurement amyloid and tau). In this group, the biomarker testing is negative/normal. In the language of the 2018 NIA-AA Research Framework, these participants have A- in their AT(N) biomarker profile, and are at clinical stage 1-3.
  Interventions: Diagnostic Test: Optical Coherence Tomography

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography — The retina is imaged using infrared light. Images collected in light are compared to those collected in darkness to extract information about function.

SUMMARY:
Years before someone experiences the symptoms of Alzheimer's disease, a compound called amyloid beta (Aβ) builds up in the brain. Excess Aβ - directly or indirectly - causes many of the symptoms of Alzheimer's dementia. However, recent studies of the FDA-approved drugs lecanemab (Leqembi®) and aducanumab (Aduhelm®) indicate that removing Aβ from the brain doesn't stop Alzheimer's. Clearly, there are other problems that need to be fixed. The investigators are interested in the cause of Aβ buildup.

Non-neuronal support cells, called glia, keep neurons healthy by regulating water and nutrient levels for the neurons. They also help clear Aβ away from neurons. Maybe Aβ builds up when glia are unhealthy.

Glia are very hard to study in the brain. Luckily, the light-sensing part of the eye - the retina - is an extension of the brain. The investigators study glia in the retina to learn about glia in the brain.

To study retinal glia, the investigators take pictures of the retina with optical coherence tomography (OCT). OCT is safe, painless, and is used in many eye clinics to look at the structure of the retina. When the investigators take OCT pictures under a bright light, and compare those to OCT pictures collected in darkness, it gives the investigators information about glial function. In a study published in 2020 ("Optical coherence tomography reveals light-dependent retinal responses in Alzheimer's disease") the investigators showed that this functional OCT measurement was different in people with Alzheimer's dementia, compared to age-matched healthy adults.

The goal of this observational study is to compare people at a pre-dementia stage of Alzheimer's disease to people who do not have any signs at all of Alzheimer's disease. By "pre-dementia stage", the investigators mean people who are either cognitively normal, or have mild cognitive impairment, but have had a medical test that shows the chemical beginnings of Alzheimer's disease. Members of the comparison group will also be cognitively normal, or have mild cognitive impairment, but had a medical test that shows utterly no signs of Alzheimer's disease.

The main question this study, is whether functional OCT can tell these two groups apart. If so, that would:

* Help build the case for glial health being important in the earliest stages of Alzheimer's, which in turn could lead to new treatment strategies, and
* Suggest that functional OCT might be used as an early (pre-dementia) screening test for Alzheimer's disease

Participants will:

* undergo a brief eye exam (the investigators will not dilate pupils for this study)
* undergo a paper-and-pencil cognitive test (to help verify "normal" or "mild cognitive impairment" status)
* take brief one-page survey to collect demographic information (like age)
* permit limited access to pre-existing medical or research records (to verify the presence/absence of the chemical beginnings of Alzheimer's disease)
* take several OCT pictures of both eyes, in light and after 2 minutes of darkness (several rounds of images are taken)

The expectation is that all study procedures will fit within 2 hours of one day.

ELIGIBILITY:
Inclusion Criteria:

* By clinician (or prior research) assessment, known to either be cognitively normal, or have mild cognitive impairment
* Known Alzheimer's biomarker status. As of 2023-JUL, this must either be an amyloid PET scan, or cerebrospinal fluid measurement of amyloid and tau levels.
* NOTE: Although this is a study of the eyes, age-typical ocular/vision complaints are permissible, so long as the the retina is thought to be healthy. This list of acceptable conditions includes most people who:

  * wear glasses
  * wear contacts
  * use over-the-counter eye drops
  * have mild cataracts (no surgery scheduled)
  * had cataracts removed
  * had eye muscle surgery (e.g., to correct eye misalignment)
  * had eyelid surgery (blepharoplasty)
  * are monitored by an ophthalmologist in case a problem with the retina develops (this is sometimes suggested for people with diabetes), but one or both retinas is/are thought to be completely healthy

Exclusion Criteria:

* Pregnant women
* Prisoners
* Known *for both eyes* to have ocular health or vision abnormalities that are not age-typical. The list of unacceptable conditions includes most people who:

  * have a special corrective lens (glasses or contact lens) prescription with a sphere greater than seven
  * currently use prescription eye drops (e.g., for glaucoma)
  * have/had prior surgical treatment for a retinal problem (e.g., retinal detachment that required surgery)
  * have/had eye injections for age-related macular degeneration

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators plan to recruit participants from:
  * Participants (or prospective participants) in research on aging and cognition at the University of California - Davis.
  * Patients (or prospective patients) of University of California - Davis neurologists.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Light-dependent Change in Optical Coherence Tomography Images | Day 1 (less than two hours)
  The investigators will obtain OCT B-scans of the span of retina between the center of the optic disc and the fovea. Each B-scan will be spatially normalized and averaged to generate a profile of retinal reflectivity versus depth into the retina. Reflectivities in light will be compared to reflectivities in darkness. In both groups, the investigators expect that (1) over the photoreceptor inner and outer segments, the retina will be more reflective in light then in darkness, (2) in the more vitread portions of the retina (the layers occupied by Müller glia), the retina will be slightly less reflective in light than in darkness.
  The investigators expect a group differences in that functional outcome. The largest group difference is expected near the exterior border of the Müller glia, where participants with a pre-dementia stage of Alzheimer's may have an exaggerated light-dependent change in reflectivity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California - Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified OCT data will be posted to a data repository.

REFERENCES:
- [Background] Bissig D, Zhou CG, Le V, Bernard JT. Optical coherence tomography reveals light-dependent retinal responses in Alzheimer's disease. Neuroimage. 2020 Oct 1;219:117022. doi: 10.1016/j.neuroimage.2020.117022. Epub 2020 Jun 5. PMID 32512126